CLINICAL TRIAL: NCT01237314
Title: Evaluation of the Glycemic Impact of Food in Patients With Type 2 Diabetes Taking Glargine and/or Exenatide
Brief Title: The Impact of Food on Blood Sugar in People With Type 2 Diabetes
Acronym: REACT2
Status: Completed | Type: Observational
Sponsor: HealthPartners Institute (Other)
Collaborators: International Diabetes Center at Park Nicollet (Other); Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: 04037-10-C
Record Dates: First submitted 2010-11-05; First posted 2010-11-09 (Estimated); Last update posted 2015-12-02 (Estimated); Status verified 2013-04

CONDITIONS: Type 2 Diabetes
Keywords: type 2 diabetes; metformin; glargine; exenatide; glycemic impact of food; continuous glucose monitoring
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- Glargine Group: After baseline titration of metformin, this group will take glargine along with metformin.
- Exenatide Group: After baseline titration of metformin, this group will take exenatide along with metformin.
- Glargine and Exenatide Group: After baseline titration of metformin, this group will take glargine and exenatide along with metformin.

SUMMARY:
This study will record the impact of food on blood glucose levels using continuous glucose monitoring (CGM).

The investigators think the impact will improve as medication doses are adjusted. The investigators also think that the impact will differ depending on the type of medication taken.

ELIGIBILITY:
Inclusion Criteria:

* Study participants who are consented for the primary study and have not yet done the baseline CGM data collection at week -2-0.

Exclusion Criteria:

* Study participants who are unable to complete the baseline CGM data collection at week -2-0.
* Study participants who are allergic to or have a food intolerance to any of the foods in the fixed meal

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Participants in Clinical Trials Study NCT01089569
Sampling Method: Non-Probability Sample
Enrollment: 46 (Actual)
Dates: Start 2010-11; Primary Completion 2013-05 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
4-hour glycemic response at 3 time points | 4 hours
  The four-hour glycemic response includes: four-hour post-meal area under the median interstitial glucose curve, post-meal interstitial glucose peak, time to peak, time to return to pre-prandial level (to within 10% of baseline with a maximum of the 4-hour post-meal fast), difference between peak and baseline, average rate of change in interstitial glucose across the 4 hour post-meal period, and percent of the 4-hour post-meal glucose readings >180 mg/dL.

CONTACTS AND LOCATIONS:
Overall Officials: Maggie Powers, PhD, Principal Investigator — International Diabetes Center at Park Nicollet; Alice Shapiro, PhD, Principal Investigator — International Diabetes Center at Park Nicollet
Locations (1):
- International Diabetes Center, Minneapolis, Minnesota, United States